CLINICAL TRIAL: NCT03597360
Title: Low Dose Ionizing Radiation Using CT Scans as a Potential Therapy for Alzheimer's Dementia (LDIR-CT-AD) Trial: A Pilot Study
Brief Title: Low Dose Ionizing Radiation Using CT Scans as a Potential Therapy for Alzheimer's Dementia: A Pilot Study
Acronym: LDIR-CT-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Jerry M Cuttler, Investigator, Baycrest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baycrest REB # 18-02
Record Dates: First submitted 2018-07-10; First posted 2018-07-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Dementia Alzheimers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CT scan subjects (Experimental): Three participants with severe Alzheimer's dementia will be studied
  Interventions: Radiation: CT scan

INTERVENTIONS:
Radiation: CT scan — Participants will receive the first LDIR treatment in one session on the same day, i.e., two CT scans of the brain that delivers a total X-ray dose (CTDIvol)10 of about 80 mGy. Participants will then be transported back to Baycrest Health Sciences. Participants will receive another LDIR treatment, i.e. a single CT scan of the brain (40 mGy), 2 weeks after the first session. They will receive a third LDIR treatment, i.e., a single CT scan of the brain (40 mGy), 2 weeks after the second session. Date, time and X-ray dose will be recorded for each participant and sent to their family physician for entry into in their health record.

SUMMARY:
The goal of this project is to determine whether low doses of ionizing radiation (LDIR) from repeat CT scanning improves function, cognition and/or behavior in severe AD.

DETAILED DESCRIPTION:
Alzheimer's dementia (AD) is a disorder of uncertain cause and pathogenesis that primarily affects older adults. It accounts for more than 50 percent of cases of dementia in the elderly and is a leading source of morbidity and mortality in the aging population. The most essential and often earliest symptom is selective memory impairment. While treatments can improve some symptoms, there is no cure or disease-modifying therapy, and the disease inevitably progresses in all patients. The mainstay of management is still symptomatic treatment of behavioral disturbances, environmental manipulations to prevent behavioural disturbances, and counseling with respect to safety issues.

The goal of this project is to determine whether low doses of ionizing radiation (LDIR) from repeat CT scanning improves function, cognition and/or behavior in severe AD. This is based upon the treatments given in 2015 to a patient in hospice in the USA with advanced AD. On July 23, she received two CT scans of her brain. Two weeks later she received a third CT scan, and two weeks after this, a fourth CT scan. She partially improved and was discharged to an Alzheimer care home.

In terms of the mechanism whereby CT scanning might lead to improvement, reactive oxygen species (ROS) are produced abundantly and constantly by aerobic metabolism in all organisms, damaging biomolecules including those in the brain. AD is postulated to be caused by the accumulation of oxidative stress damage in the brain that was not prevented, repaired or removed by the patient's own biological protective mechanisms. These systems, characterized genetically, operate against all toxins regardless of whether they are produced endogenously or by external physical, chemical or biological agents. As people age, their protection systems become progressively weaker. LDIR is postulated to stimulate adaptive protection systems. This may produce beneficial effects including improvement in AD symptoms. With about three-quarters of human tissue being water, most of the initial radiation-induced damage is radiolysis of water, producing ROS and hydrogen peroxide (H2O2). LDIR leads to mild oxidative stress and strong signaling, which up-regulates protection.The degree of stimulation likely depends upon individual genetic factors.

CT scans are approved for clinical diagnostic imaging. Approval will be requested from the Research Ethics Board (REB) at Baycrest Health Sciences and from Health Canada to use CT scanning for the experimental treatment of AD. If this pilot study is successful, i.e., if improvement is observed in the participants, then a proposal will be prepared for more comprehensive clinical studies of this novel treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with severe AD dementia (MMSE<12) between the ages of 70 to 90 years.
2. Meet the criteria of AD (NIA-AA).
3. If on any of the following medications: acetylcholinesterase inhibitors and/or memantine, participants must be on a stable dose for at least 60 days.
4. Clinically stable for at least 3 months.

Exclusion Criteria:

1. Current or past history of malignancy.
2. Previous history of radiotherapy.
3. Neurological disorder other than AD.
4. Currently receiving other experimental treatments.
5. Clinical or imaging evidence of stroke (with more than 1-2 lacunar infarcts on CT scan or MRI).
6. Major depression, bipolar affective disorder or psychosis.

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Alzheimer Disease Functional Assessment and Change Scale (ADFACS) | 20 minutes
  is a specific scale for the functional assessment of people with Alzheimer Disease. A number of specific descriptions of performance levels for each item is offered, and the caregiver is asked to identify the one that most accurately describes the patient's performance . The scale consists of 16 items for the assessment of ADL, i.e. 6 items for BADL, 10 for IADL. items are scored from 0 to 4: 0 = no impairment, 1 = mild impairment, 2 = moderate impairment, 3 = severe impairment and 4 = nonassessable, with a range from 0 to 30. BADL items are scored from 0 to 5: 0 = no impairment, 1 = mild impairment, 2 = moderate impairment, 3 = severe impairment, 4 = very severe impairment and 5 = nonassessable, with a range from 0 to 24. In each part, the 'nonassessable' answer is substituted by an estimation from the average of the responded items. The total score (IADL + BADL) ranges from 0 to 54 (from best to worst).

SECONDARY OUTCOMES:
Severe Impairment Battery (SIB) | 30 minutes
  to assess cognition
Cohen-Mansfield Agitation Index (CMAI) | 30 minutes
  The Cohen-Mansfield Agitation Index (CMAI) is a caregivers' rating questionnaire consisting of 29 agitated behaviours, each rated on a 7-point scale of frequency. It assesses the frequency of agitated behaviours in elderly persons in the long-term care setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The purpose of the information disclosure is for review by a research ethics board committee only, and is of a privileged and confidential nature.

REFERENCES:
- [Result] Ballard C, Gauthier S, Corbett A, Brayne C, Aarsland D, Jones E. Alzheimer's disease. Lancet. 2011 Mar 19;377(9770):1019-31. doi: 10.1016/S0140-6736(10)61349-9. Epub 2011 Mar 1. PMID 21371747
- [Result] Cuttler JM, Moore ER, Hosfeld VD, Nadolski DL. Treatment of Alzheimer Disease With CT Scans: A Case Report. Dose Response. 2016 Apr 1;14(2):1559325816640073. doi: 10.1177/1559325816640073. eCollection 2016 Apr-Jun. PMID 27103883
- [Result] Cuttler JM, Moore ER, Hosfeld VD, Nadolski DL. Update on a Patient With Alzheimer Disease Treated With CT Scans. Dose Response. 2017 Feb 17;15(1):1559325817693167. doi: 10.1177/1559325817693167. eCollection 2017 Jan-Mar. No abstract available. PMID 28321176
- [Result] Pollycove M, Feinendegen LE. Radiation-induced versus endogenous DNA damage: possible effect of inducible protective responses in mitigating endogenous damage. Hum Exp Toxicol. 2003 Jun;22(6):290-306; discussion 307, 315-7, 319-23. doi: 10.1191/0960327103ht365oa. PMID 12856953
- [Result] Sies H, Berndt C, Jones DP. Oxidative Stress. Annu Rev Biochem. 2017 Jun 20;86:715-748. doi: 10.1146/annurev-biochem-061516-045037. Epub 2017 Apr 24. PMID 28441057
- [Result] Feinendegen LE, Pollycove M, Neumann RD. Low-dose cancer risk modeling must recognize up-regulation of protection. Dose Response. 2009 Dec 10;8(2):227-52. doi: 10.2203/dose-response.09-035.Feinendegen. PMID 20585440
- [Result] Sies H. Hydrogen peroxide as a central redox signaling molecule in physiological oxidative stress: Oxidative eustress. Redox Biol. 2017 Apr;11:613-619. doi: 10.1016/j.redox.2016.12.035. Epub 2017 Jan 5. PMID 28110218
- [Result] Sies H, Feinendegen LE. Radiation Hormesis: The Link to Nanomolar Hydrogen Peroxide. Antioxid Redox Signal. 2017 Sep 20;27(9):596-598. doi: 10.1089/ars.2017.7233. Epub 2017 Aug 7. PMID 28699353
- [Result] Feinendegen LE, Cuttler JM. Biological Effects From Low Doses and Dose Rates of Ionizing Radiation: Science in the Service of Protecting Humans, a Synopsis. Health Phys. 2018 Jun;114(6):623-626. doi: 10.1097/HP.0000000000000833. PMID 29521814
- [Result] Manero RM, Casals-Coll M, Sanchez-Benavides G, Rodriguez-de los Reyes ON, Aguilar M, Badenes D, Molinuevo JL, Robles A, Barquero MS, Antunez C, Martinez-Parra C, Frank-Garcia A, Fernandez M, Blesa R, Pena-Casanova J; NEURONORMA Study Team. Diagnostic validity of the Alzheimer's disease functional assessment and change scale in mild cognitive impairment and mild to moderate Alzheimer's disease. Dement Geriatr Cogn Disord. 2014;37(5-6):366-75. doi: 10.1159/000350800. Epub 2014 Feb 18. PMID 24556708
- [Result] Panisset M, Roudier M, Saxton J, Boller F. Severe impairment battery. A neuropsychological test for severely demented patients. Arch Neurol. 1994 Jan;51(1):41-5. doi: 10.1001/archneur.1994.00540130067012. PMID 8274108
- [Result] Cohen-Mansfield J. Agitated behaviors in the elderly. II. Preliminary results in the cognitively deteriorated. J Am Geriatr Soc. 1986 Oct;34(10):722-7. doi: 10.1111/j.1532-5415.1986.tb04303.x. PMID 3760436
- [Result] Jack CR Jr, Albert MS, Knopman DS, McKhann GM, Sperling RA, Carrillo MC, Thies B, Phelps CH. Introduction to the recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):257-62. doi: 10.1016/j.jalz.2011.03.004. Epub 2011 Apr 21. PMID 21514247
- [Result] Sakamoto K. Radiobiological basis for cancer therapy by total or half-body irradiation. Nonlinearity Biol Toxicol Med. 2004 Oct;2(4):293-316. doi: 10.1080/15401420490900254. PMID 19330149
- [Result] Pollycove M. Radiobiological basis of low-dose irradiation in prevention and therapy of cancer. Dose Response. 2006 Nov 27;5(1):26-38. doi: 10.2203/dose-response.06-112.Pollycove. PMID 18648556
- [Result] Lemon JA, Phan N, Boreham DR. Single CT Scan Prolongs Survival by Extending Cancer Latency in Trp53 Heterozygous Mice. Radiat Res. 2017 Oct;188(4.2):505-511. doi: 10.1667/RR14576.1. Epub 2017 Jul 25. PMID 28742468
- [Result] Lemon JA, Phan N, Boreham DR. Multiple CT Scans Extend Lifespan by Delaying Cancer Progression in Cancer-Prone Mice. Radiat Res. 2017 Oct;188(4.2):495-504. doi: 10.1667/RR14575.1. Epub 2017 Jul 25. PMID 28741984